CLINICAL TRIAL: NCT01637831
Title: CPAP Therapy in Patients With Idiopathic Pulmonary Fibrosis and Obstructive Sleep Apnea. Does It Offer a Better Quality of Life and Sleep?
Brief Title: CPAP Therapy in Patients With Idiopathic Pulmonary Fibrosis and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Charalampos Mermigkis, Pulmonologist, Sleep Medicine subspecialty, University of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPAPIPF-02
Record Dates: First submitted 2012-07-04; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Obstructive Sleep Apnea; Idiopathic Pulmonary Fibrosis
Keywords: Obstructive Sleep Apnea; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Idiopathic Pulmonary Fibrosis | interventions — Continuous Positive Airway Pressure; Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with OSA and IPF (Experimental): Participants with Obstructive Sleep Apnea (OSA)and Idiopathic Pulmonary Fibrosis (IPF).This arm will complete pre-treatment questionnaires assessing sleep and quality of life, undergo six months of Continuous Positive Airway Pressure (CPAP) to treat OSA, and complete post-treatment the same questionnaires 1, 3 and 6 months later.
  Interventions: Procedure: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Procedure: Continuous Positive Airway Pressure (CPAP) — Continuous positive airway pressure (CPAP) is the gold standard for Obstructive Sleep Apnea (OSA) management. Subjects with OSA will be trained in the use of CPAP and will be instructed to use CPAP every night for 6 months. These subjects will then return for a post-treatment completion of questionnaires assessing sleep and quality of life 1, 3 and 6 months after the start of effective CPAP treatment.
  Other Names: positive pressure ventilation

SUMMARY:
The recent literature shows an increased incidence of obstructive sleep apnea (OSA) in patients with idiopathic pulmonary fibrosis (IPF). On the other hand there are no published studies related to CPAP treatment in this patient group. The investigators aim was to assess the effect of CPAP on sleep and overall life quality parameters in IPF patients with OSA and to recognize and overcome possible difficulties in CPAP initiation and acceptance by these patients.

DETAILED DESCRIPTION:
Recently published studies report a high incidence of obstructive sleep apnea (OSA) in patients with IPF. Underlying, and usually under-diagnosed OSA in these patients may be a reason for impaired sleep quality and may consequently have a negative influence on their daily activities and overall quality of life. In addition, underlying OSA may have a negative influence on the already impaired IPF-related morbidity and mortality. The absence of any effective treatment for IPF so far indicates that the recognition and treatment of generally under-diagnosed OSA in IPF patients should be a primary goal. Therefore, our primary aim in this study was to assess the results of effective CPAP therapy in terms of sleep quality and overall quality of life in IPF patients with moderate to severe OSA. The investigators used generally accepted instruments to assess quality of sleep and overall life. In addition, the investigators tried to determine and overcome the reasons for poor CPAP compliance in these patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with apnoea-hypopnoea index >15/h
* Newly diagnosed IPF

Exclusion Criteria:

* Congestive heart failure
* Chronic renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in overal quality of life parameters in IPF patients with OSA after the start of effective CPAP treatment | Day 1, Month 1, 3 and Month 6 post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sophia E Schiza, MD, PhD, Study Chair — University of Crete; Charalampos Mermigkis, MD, Study Director — Sleep Disorders Center, Pulmonary Department, 401 General Army Hospital, Athens, Greece; Izolde Bouloukaki, MD, PhD, Principal Investigator — University of Crete
Locations (1):
- Sleep Disorders Unit, Department of Thoracic Medicine, Medical School, University of Crete, Heraklion, Crete, Greece

REFERENCES:
- [Derived] Papadogiannis G, Bouloukaki I, Mermigkis C, Michelakis S, Ermidou C, Mauroudi E, Moniaki V, Tzanakis N, Antoniou KM, Schiza SE. Patients with idiopathic pulmonary fibrosis with and without obstructive sleep apnea: differences in clinical characteristics, clinical outcomes, and the effect of PAP treatment. J Clin Sleep Med. 2021 Mar 1;17(3):533-544. doi: 10.5664/jcsm.8932. PMID 33108270
- [Derived] Mermigkis C, Bouloukaki I, Antoniou KM, Mermigkis D, Psathakis K, Giannarakis I, Varouchakis G, Siafakas N, Schiza SE. CPAP therapy in patients with idiopathic pulmonary fibrosis and obstructive sleep apnea: does it offer a better quality of life and sleep? Sleep Breath. 2013 Dec;17(4):1137-43. doi: 10.1007/s11325-013-0813-8. Epub 2013 Feb 6. PMID 23386371